CLINICAL TRIAL: NCT04337944
Title: Impact of Endoscopic Assisted Anterior Hyaloid Peeling in Boston Type 1 Keratoprosthesis in Reducing Postoperative Complications
Brief Title: Endoscopic Assisted Anterior Hyaloid Peeling in Boston Type 1 Keratoprosthesis (KPro-HP-Endo)
Acronym: KPro-HP-Endo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CE19.382
Record Dates: First submitted 2020-04-03; First posted 2020-04-08 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Corneal Transplantation; Glaucoma and Ocular Hypertension; Postoperative Complications; Vitrectomy; Endoscopy
Keywords: Boston keratoprosthesis type 1; Pars plana vitrectomy; Endoscopy
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Interventional prospective study on patients receiving a Boston keratoprosthesis type 1, using a retrospective group as the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with KPro, PPV, and endoscopy (Experimental): Patients will receive at the same time a Boston keratoprosthesis type 1 (KPro) with a pars plana vitrectomy (PPV) with anterior hyaloid membrane peeling assisted by endoscopy.
  Interventions: Procedure: Boston keratoprosthesis type 1 and anterior hyaloid membrane peeling assisted by endoscopy

INTERVENTIONS:
Procedure: Boston keratoprosthesis type 1 and anterior hyaloid membrane peeling assisted by endoscopy — Patients will receive at the same time a Boston keratoprosthesis type 1 (KPro) with a pars plana vitrectomy (PPV) with anterior hyaloid membrane peeling assisted by endoscopy.

SUMMARY:
Common complications of the Boston keratoprosthesis type 1 (KPro) surgery include retroprosthetic membrane formation, glaucoma, and retinal detachment. Often pars plana vitrectomy (PPV) is performed at the same time as KPro surgery for different indications. It has been shown to reduce postoperative complications in comparison to when it is performed after the KPro surgery. Patients who receive a complete PPV with peeling of the anterior hyaloid membrane have a lower incidence of retroprosthetic membrane formation and less vision loss due to glaucoma when compared to patients with partial PPV or anterior vitrectomy. During a complete PPV, peeling of the anterior hyaloid membrane is a difficult step because visualisation is poor, but it can be improved using endoscopy. The investigators suggest that peeling of the anterior hyaloid membrane assisted by endoscopy during KPro surgery would decrease postoperative complications in comparison to a PPV done after KPro surgery and without endoscopy.

DETAILED DESCRIPTION:
Boston keratoprosthesis type 1 (KPro) surgery is the most common corneal graft and is used to restore vision in patients with high risk of failure with traditional penetrating keratoplasty. Common complications of KPro surgery include retroprosthetic membrane formation behind the backplate of the KPro. Glaucoma is the most common threat to vision rehabilitation in patients with KPro. Glaucoma is often present before surgery and progresses after KPro, seven times faster than in patients with only glaucoma. Retinal detachment is a common posterior segment complication that arises post-KPro and can lead to a serious loss of vision. Pars plana vitrectomy (PPV) is the standard treatment for patients with vitreoretinal diseases and opacities. PPV can include peeling of the anterior hyaloid membrane to ensure total resection of the vitreous body. PPV allows for example for retroprosthetic membrane excision, installation or revision of a glaucoma drainage device, or repair of retinal detachment. Often PPV is performed at the same time as KPro surgery for different indications. It has been shown to reduce postoperative complications in comparison to when it is performed after the KPro surgery. Patients who receive a complete PPV with peeling of the anterior hyaloid membrane have a lower incidence of retroprosthetic membrane formation and less vision loss due to glaucoma when compared to patients with partial PPV or anterior vitrectomy. Combined surgeries of KPro and PPV offer a complete evaluation of the optic nerve and of the retina, which would not be possible otherwise. During a complete PPV, peeling of the anterior hyaloid membrane is a difficult step because visualisation is poor, especially with a KPro in place. Visualisation can be improved using endoscopy to visualize the inside of the eye over 360 degrees. The investigators suggest that peeling of the anterior hyaloid membrane assisted by endoscopy during KPro surgery would decrease postoperative complications in comparison to a PPV done after KPro surgery and without endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 80 years old
* Informed consent
* Boston keratoprosthesis candidate
* Pars plana vitrectomy candidate
* Ability to be followed for the duration of the study

Exclusion Criteria:

* Aged less than 18 or more than 80 years old
* Inability to give informed consent
* Repeat Boston keratoprosthesis
* Repeat pars plana vitrectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Rate of retroprosthetic membrane formation | 12 months
  Rate of postoperative retroprosthetic membrane formation behind the backplate of the Boston keratoprosthesis. Retroprosthetic membrane formation is diagnosed by the investigator using an examination of the anterior chamber performed at the slit-lamp.
Rate of retinal detachment | 12 months
  Rate of postoperative retinal detachment. Retinal detachment is diagnosed by the investigator using a dilated fundus (retinal) examination performed at the slit-lamp.
Rate of glaucoma development | 12 months
  Rate of development or progression of glaucoma, determined based on intraocular pressure increase of > 21 mmHg, increase of glaucoma medications, optic nerve excavation progression, or need to undergo glaucoma filtration surgery.

SECONDARY OUTCOMES:
Proportion of patients with visual acuity better than 20/200 | 12 months
  Proportion of patients with visual acuity better than 20/200 after surgery. The visual acuity is measured using the Snellen chart.
Change of visual acuity | 12 months
  Change of visual acuity compared between before and after surgery. The visual acuity is measured using the Snellen chart.
Time to retroprosthetic membrane formation after surgery | 12 months
  Time to retroprosthetic membrane formation, calculated in months from the time of the surgery. Retroprosthetic membrane formation behind the backplate of the Boston keratoprosthesis is diagnosed by the investigator using an examination of the anterior chamber performed at the slit-lamp.
Time to retinal detachment after surgery | 12 months
  Time to retinal detachment, calculated in months from the time of the surgery. Retinal detachment is diagnosed by the investigator using a dilated fundus (retinal) examination performed at the slit-lamp.
Proportion of participants requiring glaucoma surgery | 12 months
  Proportion of participants requiring glaucoma surgery (including glaucoma drainage device, trabeculectomy or cyclophotocoagulation) after the Boston keratoprothesis surgery.
Proportion of patients with visual field loss of 30% or more | 12 months
  Proportion of patients with visual field loss of 30% or more, measured using the automated Humphrey 24-2 visual field. The loss of 30% or more of visual field is calculated using the first two postoperative tests as a reference.
Proportion of patients with thinning of the nerve fiber layer | 12 months
  Proportion of patients with thinning of the nerve fiber layer, determined by Spectral Domain Optical Coherence Tomography (SD-OCT) in average and for each of the four quadrants.
Rate of Boston keratoprosthesis complications | 12 months
  Rate of Boston keratoprosthesis complications. Complications from the Boston keratoprosthesis include: corneal melt, retroprosthetic membrane formation, retinal detachment, cystic macular edema, extrusion, hypotony, choroidal hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Harissi-Dagher, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szigiato AA, Bostan C, Nayman T, Harissi-Dagher M. Long-term visual outcomes of the Boston type I keratoprosthesis in Canada. Br J Ophthalmol. 2020 Nov;104(11):1601-1607. doi: 10.1136/bjophthalmol-2019-315345. Epub 2020 Feb 17. PMID 32066560
- [Background] Wang Q, Harissi-Dagher M. Characteristics and management of patients with Boston type 1 keratoprosthesis explantation--the University of Montreal Hospital Center experience. Am J Ophthalmol. 2014 Dec;158(6):1297-1304.e1. doi: 10.1016/j.ajo.2014.08.037. Epub 2014 Aug 28. PMID 25174898
- [Background] Harissi-Dagher M, Durr GM, Biernacki K, Sebag M, Rheaume MA. Pars plana vitrectomy through the Boston Keratoprosthesis type 1. Eye (Lond). 2013 Jun;27(6):767-9. doi: 10.1038/eye.2013.58. Epub 2013 Apr 12. PMID 23579405
- [Background] Robert MC, Pomerleau V, Harissi-Dagher M. Complications associated with Boston keratoprosthesis type 1 and glaucoma drainage devices. Br J Ophthalmol. 2013 May;97(5):573-7. doi: 10.1136/bjophthalmol-2012-302770. Epub 2013 Feb 23. PMID 23435225
- [Background] Moussally K, Harissi-Dagher M. Long-term complications associated with glaucoma drainage devices and Boston keratoprosthesis. Am J Ophthalmol. 2011 Nov;152(5):883-4; author reply 884-5. doi: 10.1016/j.ajo.2011.07.014. No abstract available. PMID 22017851
- [Background] Talajic JC, Agoumi Y, Gagne S, Moussally K, Harissi-Dagher M. Prevalence, progression, and impact of glaucoma on vision after Boston type 1 keratoprosthesis surgery. Am J Ophthalmol. 2012 Feb;153(2):267-274.e1. doi: 10.1016/j.ajo.2011.07.022. Epub 2011 Oct 7. PMID 21982110
- [Background] Dohlman CH, Zhou C, Lei F, Cade F, Regatieri CV, Crnej A, Dohlman JG, Shen LQ, Paschalis EI. Glaucoma After Corneal Trauma or Surgery-A Rapid, Inflammatory, IOP-Independent Pathway. Cornea. 2019 Dec;38(12):1589-1594. doi: 10.1097/ICO.0000000000002106. PMID 31453878
- [Background] Crnej A, Paschalis EI, Salvador-Culla B, Tauber A, Drnovsek-Olup B, Shen LQ, Dohlman CH. Glaucoma progression and role of glaucoma surgery in patients with Boston keratoprosthesis. Cornea. 2014 Apr;33(4):349-54. doi: 10.1097/ICO.0000000000000067. PMID 24531120
- [Background] Khan BF, Harissi-Dagher M, Khan DM, Dohlman CH. Advances in Boston keratoprosthesis: enhancing retention and prevention of infection and inflammation. Int Ophthalmol Clin. 2007 Spring;47(2):61-71. doi: 10.1097/IIO.0b013e318036bd8b. No abstract available. PMID 17450007
- [Background] Boscher C, Kuhn F. Endoscopic evaluation and dissection of the anterior vitreous base. Ophthalmic Res. 2015;53(2):90-9. doi: 10.1159/000370032. Epub 2015 Jan 27. PMID 25633467
- [Background] Modjtahedi BS, Eliott D. Vitreoretinal complications of the Boston Keratoprosthesis. Semin Ophthalmol. 2014 Sep-Nov;29(5-6):338-48. doi: 10.3109/08820538.2014.959204. PMID 25325859
- [Background] Yu YZ, Zou YP, Zou XL. Endoscopy-assisted vitrectomy in the anterior vitreous. Int J Ophthalmol. 2018 Mar 18;11(3):506-511. doi: 10.18240/ijo.2018.03.23. eCollection 2018. PMID 29600187